CLINICAL TRIAL: NCT02453217
Title: The Potential Efficacy and Acceptability of the Chinese Health Improvement Profile (CHIP) in Improving the Physical Health of People With Severe Mental Illness - A Pilot Clustered Randomised Controlled Trial
Brief Title: The Potential Efficacy of the Chinese Health Improvement Profile- A Pilot Clustered Randomised Controlled Trial
Acronym: CHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wai-Tong Chien (Other)
Collaborators: Castle Peak Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Wai-Tong Chien, Professor and Associate Head (Research), The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHIP1214-V1; HSEARS2014202001 (Other: Hong Kong Polytechnic University)
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Severe Mental Illness; Schizophrenia; Schizoaffective Disorder; Bipolar Affective Disorder; Cardiovascular Health
Keywords: severe mental illness; physical health screening; randomised controlled trial; health behaviour change
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chinese CHIP (Experimental): Chinese Health Improvement Profile (CHIP) screening and intervention
  Interventions: Behavioral: Chinese CHIP; Other: Treatment as usual
- Treatment as usual (No Intervention): Routine community mental health care and medical outpatient appointments

INTERVENTIONS:
Behavioral: Chinese CHIP — The CHIP physical health screening tool will be used by community psychiatric nurses in the treatment group to assess patients' physical health risk and identify problematic lifestyle behaviours. The findings from the assessment will be used to devise an individualized care plan with patients. This treatment plan may involve community psychiatric nurses collaborated with psychiatrists, drawing patients attention to indicators of physical health risk by using a traffic light system The community nurses will use motivational interviewing approaches to make patients be aware of their physical health risks and enhance their motivation to adopt healthier behaviours.
  Other Names: CHIP
  Arms: Chinese CHIP
Other: Treatment as usual — The routine community mental health care provided by the community psychiatric nursing service and outpatient clinic.
  Other Names: TAU
  Arms: Chinese CHIP

SUMMARY:
The investigators programme of research will evaluate an existing physical health care screening intervention with the aim of helping Community Psychiatric Nurses (CPN) to improve the physical health wellbeing of people with a SMI.

This pilot clustered randomised controlled trial aims to establish the potential efficacy and acceptability of the Chinese Health Improvement Profile (CHIP) in improving the physical health of people with severe mental illness.

DETAILED DESCRIPTION:
This pilot study will use a non-blinded parallel group clustered randomised controlled trial design.

The study will be carried out by CPNs with community-dwelling people aged 18-65 who have a psychiatric diagnosis of SMI (i.e. schizophrenia, schizoaffective disorder, other psychotic disorder or bipolar affective disorder) and at the point of recruitment are being treated in the community. It will investigate the potential clinical impact of the use of the CHIP tool when used by CPNs with this patient group. Because the CHIP is designed to be used as both an enhanced physical health risk screening tool and as an instrument to direct appropriate clinical interventions the investigators will ask the patients' allocated CPNs to recruit consenting patients , collect outcome measure data and where appropriate use the CHIP tool with patients that they work with within their routine clinical practice.

Primary objective:

To test the potential efficacy and acceptability of the CHIP intervention compared to treatment as usual on patients' physical well- being over a 12 month period.

Secondary objectives:

To measure and compare changes in perceived mental well-being between the groups as measured at baseline, and at 6 months and 12 months after the start of the intervention.

To establish differences in the objective physical health state of patients between the groups at 12 months as indicated by data routinely recorded in medical/outpatient/nursing notes during the duration of study.

To establish changes in health behaviours and physical indicators of cardiovascular risk within the intervention group between baseline and 12 months after the start of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Those psychiatric outpatients under the care of the community psychiatric nursing service who are:

* Aged 18-65 years;
* Having a case-note diagnosis (as confirmed by a registered clinician) within the illness group entitled "severe mental illness" (SMI) containing schizophrenia, schizoaffective disorder, other psychotic disorders, depressive or bipolar affective disorder (type 1 or 2); and
* Able to speak Chinese/English
* Able to provide written informed consent and considered safe and competent to participate in the study (as suggested by attending psychiatrist).

Exclusion Criteria:

* Co-morbidity of learning disability or organic brain diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Self-reported physical well being | 6 months after intervention
  The primary outcome will be measured using the widely used and well-established Chinese version of the physical and mental health measure (SF12v2-PCS-12 subscale).
Self-reported physical well being | 12 months after intervention
  The primary outcome will be measured using the widely used and well-established Chinese version of the physical and mental health measure (SF12v2-PCS-12 subscale).

SECONDARY OUTCOMES:
Self-reported mental health | 6 months after intervention
  The perceived mental health will be measured using the widely used and well-established Chinese version of the physical and mental health measure (SF12v2-MCS-12 subscale).
Satisfaction with services | 12 months after intervention
  Patients' satisfaction with the services received will be measured with the Chinese language version of the Client Satisfaction Questionnaire (CSQ8)
Self-reported mental health | 12 months after intervention
  The perceived mental health will be measured using the widely used and well-established Chinese version of the SF12v2 (MCS-12 subscale).

OTHER OUTCOMES:
The Chinese CHIP data (treatment group only) | 12 months after intervention
  The data recorded from the individual items of the CHIP will be compared between baseline and at 12 months after the start of the intervention.
Physical state | 12 months after intervention
  The data relating to patients' physical state that are routinely recorded in medical, outpatient and nursing notes during study period will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Bressington, PhD, Principal Investigator — The Hong Kong Polytechnic University; Wai Tong Chien, PhD, Study Director — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware, J.E., Jr., Kosinski, M., Dewey, J.E. How to Score Version 2 of the SF-36® Health Survey (Standard & Acute Forms). Lincoln, RI: QualityMetric Incorporated, 2000.
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] White J, Gray R, Jones M. The development of the serious mental illness physical Health Improvement Profile. J Psychiatr Ment Health Nurs. 2009 Jun;16(5):493-8. doi: 10.1111/j.1365-2850.2009.01375.x. Epub 2008 Mar 9. PMID 19538607
- [Result] Bressington D, Mui J, Yu C, Leung SF, Cheung K, Wu CST, Bollard M, Chien WT. Feasibility of a group-based laughter yoga intervention as an adjunctive treatment for residual symptoms of depression, anxiety and stress in people with depression. J Affect Disord. 2019 Apr 1;248:42-51. doi: 10.1016/j.jad.2019.01.030. Epub 2019 Jan 28. PMID 30711868
- [Result] Bressington D, Yu C, Wong W, Ng TC, Chien WT. The effects of group-based Laughter Yoga interventions on mental health in adults: A systematic review. J Psychiatr Ment Health Nurs. 2018 Oct;25(8):517-527. doi: 10.1111/jpm.12491. PMID 30030938
- [Derived] Bressington D, Mui J, Tse ML, Gray R, Cheung EF, Chien WT. Cardiometabolic health, prescribed antipsychotics and health-related quality of life in people with schizophrenia-spectrum disorders: a cross-sectional study. BMC Psychiatry. 2016 Nov 18;16(1):411. doi: 10.1186/s12888-016-1121-1. PMID 27863522